CLINICAL TRIAL: NCT05363748
Title: A Prospective Study of the Renal Artery Fibromuscular Dysplasia Registry in China
Brief Title: Renal Artery Fibromuscular Dysplasia Registry
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji-Guang Wang, Director of the Shanghai Institute of Hypertension and the Department of Hypertension, Shanghai Jiao Tong University School of Medicine
Other Study IDs: RA-FMD
Record Dates: First submitted 2022-04-01; First posted 2022-05-06 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Renal Artery Fibromuscular Dysplasia
Keywords: Renal Artery Fibromuscular Dysplasia; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Patients with renal artery FMD will be asked for at least collection of an EDTA sample for DNA extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation group: sequential

SUMMARY:
1. Study name: A Prospective Study of the Renal artery fibromuscular dysplasia Registry in China
2. Rationale: Fibromuscular dysplasia (FMD) is an idiopathic systemic noninflammatory arterial disease resulting in narrowing of medium-sized arteries. Renal arteries are most commonly involved vessels, although it can also affect arteries in other vascular territories. Renal artery FMD is the second frequent cause of renovascular hypertension , especially in adolescents. The pathogenesis of FMD is still not understood. There were little Asians in the United States and the European/International FMD registry.
3. Objective: 1) To describe the characteristics of renal artery FMD; 2) To identify environmental/ hormonal factors and exposures (for example smoking) associated with the onset and progression of renal artery FMD; 3)To identify baseline characteristics of the disease associated with an increased risk of complications such as dissections, aneurysms, stroke or myocardial infarction; 4) To provide evidence-based algorithms for the management and follow-up of patients with renal artery FMD; 5) To establish a comprehensive imaging resource including a wide range of presentations of renal artery FMD.
4. Study design: Prospective, multi-center, observational study.
5. Study population: renal artery fibromuscular dysplasia
6. Data Collections: 1) Data on demographic characteristics, clinical characteristics, blood routine, biochemical and plasmic electrolytes and vascular imaging were collected using a questionnaire; 2) The diagnosis of renal artery FMD was based on the identification of focal or multifocal FMD lesions in at least one arterial bed by computed tomography angiography, magnetic resonance angiography and/or digital subtraction angiographies; 3) For the patients with renal artery FMD, screening was performed to assess most arteries and multivessel FMD would be collected; 4) All patients would be followed up.
7. Treatment: Standardized diagnosis and treatment procedure as recommended in the International Consensus on the diagnosis and management of fibromuscular dysplasia.
8. Follow up: 3, 6, 12 months after diagnosis and every year after enrolled.
9. Sample size estimation: About 5 hundred.
10. Timeline: Start of subjects' enrollment: Jan 2021; End of subjects enrollment: December 2026; End of study: December 2036.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

DETAILED DESCRIPTION:
1. Study name: A Prospective Study of the Renal artery fibromuscular dysplasia Registry in China
2. Rationale: Fibromuscular dysplasia (FMD) is an idiopathic systemic noninflammatory arterial disease resulting in narrowing of medium-sized arteries and causes stenosis, aneurysm, occlusion, or dissection. Renal arteries are most commonly involved vessels, although it can also affect arteries in other vascular territories. Renal artery FMD is the second frequent cause of renovascular hypertension (RVH), especially in adolescents. FMD often affects two or more arterial beds (prevalence of multivessel FMD: 57 to 66%). Despite traditional views on the role of female hormones, mechanical factors and, more recently, smoking, the pathophysiology of FMD is still not well understood. There were little Asians in the United States and the European/International FMD registry.
3. Objective: 1) To describe the characteristics of renal artery FMD in men and women, older and younger patients and according to different arterial manifestations, ethnic origin in order to individualize management and prevent complications; 2) To identify environmental/ hormonal factors and exposures (for example smoking) associated with the onset and progression of renal artery FMD;3)To identify baseline characteristics of the disease associated with an increased risk of complications such as dissections, aneurysms, stroke or myocardial infarction; 4) To provide evidence-based algorithms for the optimal management and follow-up of patients with renal artery FMD; 5) To establish a comprehensive imaging resource including a wide range of presentations of renal artery FMD, which may be used to improve knowledge and raise awareness in the medical community.
4. Study design: Prospective, multi-center, observational study.
5. Study population: patients with renal artery fibromuscular dysplasia who signed the informed consent will be eligible. The following patients are eligible for inclusion: 1) Patients with established renal artery FMD, at least one string-of-beads (multifocal FMD) or focal stenosis (focal FMD). 2) Patients with so-called "atypical FMD" or "FMD-like presentation", i.e. patients presenting with at least one dissection or 2 aneurysms < 60-year-old, in the absence string-of-beads, focal stenosis or evidence of inherited arteriopathy. 3) Children with renal artery FMD may be also included, provided they meet the inclusion criteria and there is no evidence of underlying syndromes such as Williams syndrome, Alagille syndrome or type 1 Neurofibromatosis.
6. Data Collections: 1) Data on demographic characteristics (age, gender, height, and ethnicity), clinical characteristics [seated office systolic and diastolic blood pressure (BP), smoking, family history on hypertension or FMD, concomitant diseases, current medications, age at diagnosis of renal artery FMD, angiographic subtype of renal artery FMD, symptoms of renal artery FMD at diagnosis and associated atheroma lesions], blood routine, biochemical and plasmic electrolytes and vascular imaging (arterial beds explored, imaging modality, type, and site of lesions for each vascular bed) were collected using a questionnaire; 2) The diagnosis of renal artery FMD was based on the identification of focal or multifocal FMD lesions in at least one arterial bed by computed tomography angiography (CTA), magnetic resonance angiography(MRA) and/or digital subtraction angiographies (DSA), as recommended in the first international FMD Consensus; 3) For the patients with renal artery FMD, screening was performed to assess all arteries (for example: cerebrovascular, mesenteric, aorta, renal, coronary, visceral, upper and lower extremity arteries) and multivessel FMD would be collected. 4) All patients would be followed up and data ( for example: the blood pressure and restenosis) would be evaluated again.
7. Treatment: Standardized diagnosis and treatment procedure as recommended in the International Consensus on the diagnosis and management of fibromuscular dysplasia.
8. Follow up: 3, 6, 12 months after diagnosis and every year after enrolled.
9. Sample size estimation: About 5 hundred.
10. Timeline: Start of subjects' enrollment: Jan 2021; End of subjects enrollment: December 2026; End of study: December 2036.
11. Organization: The Centre for Epidemiological Studies and Clinical Trials, Ruijin Hospital, Shanghai, China.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent;
2. Patients diagnosed with renal artery fibromuscular dysplasia (FMD), i.e. at least one string-of-beads (multifocal FMD) or focal stenosis (focal FMD). The diagnosis needs to be confirmed by at least one of the following imaging modalities: CT-angiography, MR-angiography or catheter-based angiography;
3. Patients with so-called "atypical renal artery FMD" or "renal artery FMD-like presentation", i.e. patients presenting with at least one dissection or 2 aneurysms < 60-year-old, in the absence string-of-beads, focal stenosis or evidence of inherited arteriopathy;
4. Patients with established renal artery FMD younger than 18 years, without evidence of underlying syndromes such as Williams syndrome, Alagille syndrome or type 1 Neurofibromatosis;

Exclusion Criteria:

1. Not eligible for inclusion or in situations considered unqualified for the study by the investigator;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with renal artery fibromuscular dysplasia who signed the informed consent will be eligible. The following patients are eligible for inclusion: 1) Patients with established renal artery FMD, at least one string-of-beads (multifocal FMD) or focal stenosis (focal FMD). 2) Patients with so-called "atypical FMD" or "FMD-like presentation", i.e. patients presenting with at least one dissection or 2 aneurysms < 60-year-old, in the absence string-of-beads, focal stenosis or evidence of inherited arteriopathy. 3) Children with renal artery FMD may be also included, provided they meet the inclusion criteria and there is no evidence of underlying syndromes such as Williams syndrome, Alagille syndrome or type 1 Neurofibromatosis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2036-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of focal or multifocal FMD | 1 day
  The percentage of focal or multifocal subtype in the renal artery FMD in China
The percentage of multivessel FMD in the renal artery FMD | 1 week
  The percentage of multivessel FMD in the renal artery FMD in China
The change of blood pressure | 10 years
  Comparison of blood pressure between baseline and 3/6/12 months (every year) after percutaneous transluminal angioplasty.
The rate of restenosis of renal artery FMD | 10 years
  The rate of restenosis of renal artery FMD after percutaneous transluminal angioplasty
The rate of incidence of cardiovascular events | 10 years
  The rate of incidence of cardiovascular events in the renal artery FMD patients, such as cerebral infarction, hypertensive nephropathy, myocardial infarction and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Jiguang Wang, PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Locations (1):
- Shanghai Institite of Hypertension, Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided